CLINICAL TRIAL: NCT00715468
Title: Prospective, 6 Month, Open Label, Conversion Study From MMF to MYFORTIC* Evaluating the Severity of GI Symptoms and MPA Metabolite as a Surrogate Marker of MYFORTIC
Brief Title: Prospective, 6 Month, Open Label, Conversion Study From Mycophenolate Mofetil (MMF) to PRMYFORTIC*
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Suzon Collette, Transplantation Nephrologist, Maisonneuve-Rosemont Hospital
Other Study IDs: CERL080ACA07
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Late Complication From Kidney Transplant

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Treatment with MMF often results in adverse GI events, which can lead to dose reductions of MMF and decreased graft function. Enteric-coated mycophenolate sodium (MYFORTIC*) was developed as an alternative formulation of MPA to improve upper GI tract side effects. An improvement in the severity of GI side effects could result in an increased tolerance to MPA and an improvement in patient quality of life. This study will use the GSRS to evaluate improvement in gastrointestinal symptoms.

DETAILED DESCRIPTION:
This study will evaluate the change in the total gastrointestinal symptom rating scale (GSRS) score at baseline versus month 1,at baseline versus month 3 and at baseline versus month 6 after conversion from MMF to PRMYFORTIC* .

ELIGIBILITY:
Inclusion Criteria:

* Received a kidney transplant at least six months
* stable graft function (no increased creatinine > 20% in the previous 4 weeks)
* Receiving immunosuppressive regimen with stable dose of MMF for at least 4 weeks
* Immunosuppressive regimen with a dose of MMF (dose≤ 2.0 g/day) at least 4 weeks OR C0 MMF < 1.4 µg/ml at visit 1 OR patients receiving MMF who have GI side effects
* Willing to provide written informed consent
* Women of childbearing age must have a negative pregnancy test and use a medically acceptable method of contraception throughout the treatment period;
* Over 18 years of age.

Exclusion Criteria:

* GI symptoms assumed or known not to be caused by MPA therapy;
* Acute rejection episode ≤ 4 weeks prior to study enrollment;
* Liver disease interfering with enterohepatic recirculation, such as active hepatitis B, active hepatitis C, autoimmune hepatitis and liver cirrhosis;
* Female patients who are pregnant, lactating or of child bearing potential and not practicing an approved method of birth control;
* Active bacterial, viral or fungal infection;
* Presence of psychiatric illness that in the view of the investigator would interfere with study requirements;
* Known sensitivity to the study drug;
* Receiving any investigational drug or have received any investigational drug within 30 days prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: renal transplant patients who have received a transplant at least 3 months and experiencing Gastrointestinal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2007-08; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in the total gastrointestinal symptom rating scale(GSRS) score at baseline vs 1 month, va 3 month and vs 6 month | 1 month- 3 month-6 month

SECONDARY OUTCOMES:
evaluate the change in the diarrhea GSRS subscale on a per patient basis | at month 6
incidence of adverse events and serious events at months 3 an d6 will be evaluated | month 3 and 6
Renal function and incidence of acute rejection | 1-3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Suzon Collette, Md, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada